CLINICAL TRIAL: NCT04326855
Title: Methodological Validation of an Intermittent Shuttle Walking Protocol in the Context of Pulmonary Rehabilitation in Patients With Advanced COPD
Brief Title: Validation of an Intermittent Shuttle Walking Protocol in Patients With COPD
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northumbria University (Other)
Collaborators: Royal Victoria Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 280032
Record Dates: First submitted 2020-03-02; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Chronic Obstructive Lung Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: This is a cross sectional interventional trial. The same group of COPD patients will perform four shuttle walking protocols. The intermittent shuttle walking protocol will be compared to the endurance shuttle walking protocol (control) which is commonly implemented in the PR settings. The intermittent shuttle walking protocol will be performed twice by all patients to obtain test re-test reliability in terms of distance walked, of cardiorespiratory and symptoms responses. The order of testing will be determined by balanced sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 patients with advanced COPD (Experimental): This will be a cross sectional observational study. COPD patients will be recruited from those referred to the Pulmonary Rehabilitation programme at RVI Hospital in Newcastle upon Tyne. Potentially eligible patients will be identified by the physiotherapy team within the Trust, who will provide initial information about the study. Delegated investigators will confirm eligibility and discuss full details of the trial. Patients will be given time to consider participation in the trial before written informed consent is obtained.
  Interventions: Other: Incremental shuttle walking protocol (ISWT); Other: Endurance shuttle walking (ESW) protocol; Other: First Intermittent shuttle walking protocol; Other: Second Intermittent shuttle walking protocol; Other: Focus group study

INTERVENTIONS:
Other: Incremental shuttle walking protocol (ISWT) — Patients will perform an incremental shuttle walk test to the limit of tolerance to establish peak walking speed. The test will be developed in a 10-m course corridor, and it will be externally-paced via a recorded metronome that gives a signal for each stride. The walking pace will be increased every minute and the test will be terminated when the individual is no longer able to keep up the pace. Pulmonary variables will be recorded breath-by-breath. Cardiac output will be assessed every min. Arterial oxygen saturation will be measured by a pulse oximeter. Patients will score the intensity of their breathlessness and leg discomfort using the 1-10 Borg's scale every minute.
Other: Endurance shuttle walking (ESW) protocol — Subsequently, during the second visit all patients will perform the continuous endurance shuttle walk (ESW) protocol to the limit of tolerance at a walking speed corresponding to 85% of VO2 peak derived by the ISWT (visit 1). During the ESW protocol patients will receive standardized instructions to walk for as long as possible although there will be a predetermined 6 minute maximum point. No further encouragement will be provided during the exercise performance. The test will be terminated when the individual is no longer able to keep up the pace or stops due to intolerable exertional symptoms. Gas exchange and cardiorespiratory variables will be assessed as per visit 1.
Other: First Intermittent shuttle walking protocol — All patients will perform an intermittent shuttle walking protocols to the limit of tolerance (visit 3) by alternating 1-min walking bouts sustained at a walking speed equivalent to 85% peak (equivalent to the continuous ESW protocol) with 1-min rest periods.The test will be terminated when the individual is no longer able to keep up the pace or stops due to intolerable exertional symptoms although there will be a predetermined 20 minute maximum point.Gas exchange and cardiorespiratory variables will be assessed as per visit 1.
Other: Second Intermittent shuttle walking protocol — To obtain test re-test reliability in terms of distance walked, of cardiorespiratory and symptoms responses this intermittent shuttle walking protocol will be repeated on a different day (visit 4). The test will be terminated when the individual is no longer able to keep up the pace or stops due to intolerable exertional symptoms although there will be a predetermined 20 minute maximum point. Gas exchange and cardiorespiratory variables will be assessed as per visit 1.
  Other Names: Test-retest reliability study
Other: Focus group study — Semi-structured interviews to explore patients' preferences of undertaking the intermittent or continuous ESW protocols and healthcare professionals' perceived factors affecting the implementation of these protocols in the PR setting. These semi-structured interviews consist of questions in some degree predetermined order but still ensures flexibility in the way issues are addressed to the patients. Conversation is sustained in an informal tone and lasts for about an hour. Participants are allowed for an open response in their own words.
  Other Names: Semi-structured Interviews

SUMMARY:
In the UK, field-based walking is prescribed in the pulmonary rehabilitation (PR) setting as a convenient, less resource-intensive, and highly responsive exercise modality in COPD patients. However, endurance time during the implementation of field-based walking protocols, such as the endurance shuttle walking (ESW) protocol, is limited to only a few minutes secondary to intense exertional symptoms. It therefore seems sensible to develop an intermittent field-based walking protocol that would prolong endurance time and walking distance compared to the commonly implemented in the PR setting continuous ESW protocol. The aim of this study is three-fold: 1) to identify whether an intermittent shuttle walking protocol significantly prolongs walking distance compared to the widely implemented continuous ESW protocol in the PR setting in patients with advanced COPD; 2) to investigate the test re-test reliability of the distance walked during the intermittent shuttle walking protocol; and 3) to explore patients' and health care professionals' experiences of implementing the intermittent walking protocol and the perceived factors affecting the implementation of these protocols in the PR setting.

The study hypothesis is that the intermittent shuttle walking protocol would be associated with lower dynamic hyperinflation and breathlessness, thereby facilitating an increase in walking distance compared to the continuous ESW protocol.

The same group of patients with advanced COPD will initially perform an incremental shuttle walk test (ISWT) (visit 1) to establish peak walking speed and subsequently patients will perform the continuous ESW protocol (visit 2) at a walking speed corresponding to 85% of peak walking speed to the limit of tolerance. On two additional visits (visits 3 and 4) patients will perform two intermittent shuttle walking protocols to the limit of tolerance by alternating 1-min walking bouts at a walking speed corresponding to 85% peak walking speed (equivalent to the ESW protocol) with 1-min rest periods in between walking bouts to establish the reproducibility of this protocol. Focus group interviews with patients and healthcare professionals will be conducted to explore perceptions of undertaking and implementing, respectively the intermittent walking protocol.

DETAILED DESCRIPTION:
Although previous research in the area of pulmonary rehabilitation in COPD has documented that high intensity exercise induces greater benefits than moderate intensity exercise, patients with advanced COPD patients cannot sustain sufficiently high intensities for long periods of time due to exertional breathlessness. While patients are limited by breathlessness during continuous modes of exercise, intermittent exercise is considered to be a good alternative strategy for patients with advanced COPD as it is associated with reduced exertional symptoms. Intermittent exercise consists of repeated brief bouts of physical activity at a high intensity alternated with short periods of recovery. The rationale for the implementation of intermittent exercise in healthy people and athletes has been the capacity to impose high loads to peripheral muscles without overloading the cardiorespiratory system. Working at high intensities with limited exertional symptoms enables severe COPD patients to achieve greater exercise volumes and in extend greater peripheral muscle adaptations, thereby improving exercise tolerance. International (ATS/ERS) and national (BTS) position statements for pulmonary rehabilitation recommend intermittent exercise for patients with advanced COPD. Despite the well-documented benefits of intermittent exercise, very few pulmonary rehabilitation centres in the UK employ this modality. The reason is that most of the community-based pulmonary rehabilitation programmes lack of infrastructure (stationary cycle ergometers, treadmills, rowing machines, etc.) and healthcare professionals to implement interval exercise. Hence, it is necessary to develop alternative, easily implemented and affordable, in terms of symptoms, exercise particularly for patients with advanced COPD across the community- and hospital- based pulmonary rehabilitation setting in the UK.

In the UK, field-based walking training is prescribed in the PR setting as a convenient, less resource-intensive, and highly responsive exercise modality in patients with COPD. However, in 2018, the National COPD Audit Report, reported that only 62% of enrolled patients completed a PR programme, highlighting significant drop-out rates (38%) between initial assessment and programme completion. Intense exertional symptoms during the prescribed exercise regimes was the main identified factor responsible for non-completion rates. In 1999, Revill et al, introduced a standardized, externally-paced (continuous) endurance shuttle walk (ESW) protocol as a highly responsive and repeatable assessment tool to measure endurance capacity. The ESW protocol sustained at a relatively high intensity (85% peak walking speed derived by the Incremental Shuttle Walk Test - ISWT) is commonly employed today as a walking training modality in the PR setting across the UK. However, endurance time during implementation of ESW protocol is limited to only a few minutes (5-8 minutes) secondary to intense exertional symptoms. In particular, both breathlessness and leg discomfort are considered to limit endurance time during the ESW protocol, thus suggesting that it is a highly physically demanding task for advanced COPD patients.

It therefore seems sensible to develop an intermittent shuttle walking protocol imposing sufficiently intense loads to the cardiorespiratory system and the locomotor muscles without inducing intense exertional symptoms. In turn, this would prolong endurance time and walking distance compared to the commonly implemented continuous ESW protocol. It is envisaged that an intermittent walking protocol for patients with advanced COPD will facilitate participation and successful completion of a PR programme.

Research Aims

1. To identify whether an intermittent shuttle walking protocol is associated with tolerable exertional symptoms, thereby prolonging walking distance compared to the widely implemented continuous ESW protocol in the PR settings for patients with advanced COPD.
2. To investigate the reproducibility of the distance walked during the intermittent shuttle walking protocol.
3. To explore both patients' and health care professionals' experiences of undertaking and implementing, respectively the intermittent shuttle walking and the perceived factors affecting the implementation of this protocol in the PR setting.

Research Objectives

1. To compare walking distance, cardiorespiratory and symptom responses (breathlessness and leg discomfort) of an intermittent shuttle walking protocol (sustained at 85% of peak walking speed) to the commonly applied continuous ESW protocol (also sustained at 85% of peak walking speed) in the PR setting.
2. To evaluate the test-retest reliability of distance walked, cardiorespiratory and symptom responses during the intermittent shuttle walking protocols.
3. To explore patients' preferences of undertaking an intermittent shuttle walking protocol, and the health care professionals' perceived barriers and facilitators affecting the implementation of this protocol in the pulmonary rehabilitation setting.

Study Design

1. A cross sectional observational study to compare distance walked, cardiorespiratory responses and symptoms of patients undertaking two shuttle walking protocols, namely the continuous endurance shuttle walking (ESW) and the intermittent shuttle walking protocol.
2. A test-retest reliability study to evaluate the validity of the intermittent shuttle walking protocol in terms of walking distance, cardiorespiratory responses and symptoms.
3. A qualitative focus group study to explore patients' preferences of undertaking the intermittent or continuous ESW protocols and healthcare professionals' perceived factors affecting the implementation of these protocols in the PR setting.

Study population

COPD patients will be recruited from those referred to the Pulmonary Rehabilitation programme at RVI Hospital in Newcastle upon Tyne. Potentially eligible patients will be identified by the physiotherapy team within the Trust, who will provide initial information about the study. Delegated investigators will confirm eligibility and discuss full details of the trial. Patients will be given time to consider participation in the trial before written informed consent is obtained.

Planned Interventions

Following confirmation of eligibility, informed consent and baseline lung assessment, all patients will be asked initially during the first visit to perform an incremental shuttle walk test (ISWT) to the limit of tolerance to establish peak walking speed without prior practice. The test will be developed in a 10-m course corridor, and it will be externally-paced via a recorded metronome that gives a signal for each stride. The walking pace will be increased every minute and the test will be terminated when the individual is no longer able to keep up the pace or stops due to intolerable exertional symptoms.

Subsequently, during the second visit all patients will perform the continuous endurance shuttle walk protocol (ESW) to the limit of tolerance at 85% peak walking speed derived by the ISWT (visit 1). During the ESW protocol patients will receive standardized instructions to walk for as long as possible. No further encouragement will be provided during the exercise performance. The test will be terminated when the individual is no longer able to keep up the pace or stops due to intolerable exertional symptoms.

Following completion of the ESW protocol, patients will perform on two different days two intermittent shuttle walking protocols to the limit of tolerance (visits 3 & 4) by alternating 1-min walking bouts sustained at a walking speed equivalent to 85% peak (equivalent to the continuous ESW protocol) with 1-min rest periods. To obtain test re-test reliability in terms of distance walked, of cardiorespiratory and symptoms responses this intermittent shuttle walking protocol will be repeated in visit 4 (Diagram 4). The test will be terminated when the individual is no longer able to keep up the pace or stops due to intolerable exertional symptoms.

Throughout the ISWT, the ESW and the two intermittent protocols, pulmonary gas exchange and ventilatory variables will be recorded breath-by-breath (K4b2, Cosmed,). Cardiac output, stroke volume and heart rate will be assessed by a portable cardio-impedance cardiography system (Physio flow, Manatec). Percentage arterial oxygen saturation (SpO2) will be measured by a pulse oximeter. Throughout testing, changes in operational lung volumes will be dynamically evaluated by performing inspiratory capacity (IC) manoeuvres. Patients will score the intensity of their breathlessness and leg discomfort using the 1-10 Borg's scale every minute during the ESW and the intermittent walking protocols.

3. Qualitative focus group study (semi-structured interviews)

Study Outcomes:

The primary outcome is the distance walked (in meters) during the intermittent shuttle walking protocol compared to the widely implemented continuous ESW protocol in the PR setting for patients with advanced COPD.

Secondary Outcomes:

* Cardiorespiratory responses (ventilatory and circulatory responses)
* Exertional Symptoms (breathlessness and leg discomfort)
* Acceptability and feasibility (assessed by semi-structured interviews)

Sample Size Calculation

The calculation is based on the minimal important difference estimates (MID) of 82 (m) of the ESW protocol and the standard deviation (SD) of 113 (m) between the different performances of ESW walked distance improvement from the same study. Using an alpha significance level of 0.05 (2-sided) and 80% power, a minimum sample size of 17 was calculated to be sufficient. To compensate for possible drop-outs (i.e. 20%) across the different assessment points over a period of 12 months, 20 patients will be recruited to allow the allocation of the different protocols with ordered sequence across the group of COPD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 40 years or older.
2. Current or previous smoking history: 10 or more pack years.

Exclusion Criteria:

1. Orthopaedic, neurological or other concomitant diseases that significantly impair normal biomechanical movement patterns, as judged by the investigator.
2. Moderate or severe COPD exacerbation within 6 weeks.
3. Unstable cardiac arrhythmia.
4. Unstable ischaemic heart disease, including myocardial infarction within 6 weeks.
5. Moderate or severe aortic stenosis or hypertrophic obstructive cardiomyopathy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Walking distance | The intervention will be performed within 30 days from the date of patient recruitment. Outcome 1 will be assessed at the 20th minute for the intermittent walking protocol.
  Distance walked during the intermittent shuttle walking protocol compared to the distance walked during the continuous endurance shuttle walking protocol assessed in meters.
  Change in walking distance covered during the intermittent walking protocol.

SECONDARY OUTCOMES:
Change in Peak oxygen consumption (VO2 peak) | The intervention will be performed within 30 days from the date of patient recruitment.Outcome 2 will be assessed at the 20th minute for the intermittent walking protocol.
  Oxygen consumption will be monitored breath-by-breath with a portable telemetric system. Change in Oxygen consumption will be assessed at the end of the intermittent walking protocol.
Change in Cardiac output | The intervention will be performed within 30 days from the date of patient recruitment.Outcome 3 will be assessed at the 20th minute for the intermittent walking protocol.
  Cardiac output responses will be assessed non-invasively by cardio impedance technology.
  Change in cardiac output will be measured at the end of the intermittent walking protocol.
Change in Exertional Symptoms (breathlessness and leg discomfort) | The intervention will be performed within 30 days from the date of patient recruitment.Outcome 4 will be assessed at the 20th minute for the intermittent walking protocol.
  Change in breathlessness and leg discomfort will be assessed by mentioning a number in Borg's scale (lowest:1-highest: 10) and will be scored at the 20th minute for the intermittent walking protocol.
Change in Minute Ventilation | The intervention will be performed within 30 days from the date of patient recruitment.Outcome 5 will be assessed at the 20th minute for the intermittent walking protocol.
  Minute Ventilation will be monitored breath-by-breath with a portable telemetric system.
  Change in Minute ventilation will be assessed at the end of the intermittent walking protocol.
Change in Inspiratory Capacity | The intervention will be performed within 30 days from the date of patient recruitment. Outcome 6 will be assessed at the 20th minute for the intermittent walking protocol.
  Inspiratory Capacity manoeuvres will be performed and monitored with a portable telemetric system.
  Change in inspiratory capacity will be assessed at the end of the intermittent walking protocol.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kruis AL, Smidt N, Assendelft WJ, Gussekloo J, Boland MR, Rutten-van Molken M, Chavannes NH. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2013 Oct 10;(10):CD009437. doi: 10.1002/14651858.CD009437.pub2. PMID 24108523
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Vogiatzis I, Zakynthinos S. Factors limiting exercise tolerance in chronic lung diseases. Compr Physiol. 2012 Jul;2(3):1779-817. doi: 10.1002/cphy.c110015. PMID 23723024
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Bolton CE, Bevan-Smith EF, Blakey JD, Crowe P, Elkin SL, Garrod R, Greening NJ, Heslop K, Hull JH, Man WD, Morgan MD, Proud D, Roberts CM, Sewell L, Singh SJ, Walker PP, Walmsley S; British Thoracic Society Pulmonary Rehabilitation Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guideline on pulmonary rehabilitation in adults. Thorax. 2013 Sep;68 Suppl 2:ii1-30. doi: 10.1136/thoraxjnl-2013-203808. No abstract available. PMID 23880483
- [Background] Spruit MA, Pitta F, Garvey C, ZuWallack RL, Roberts CM, Collins EG, Goldstein R, McNamara R, Surpas P, Atsuyoshi K, Lopez-Campos JL, Vogiatzis I, Williams JE, Lareau S, Brooks D, Troosters T, Singh SJ, Hartl S, Clini EM, Wouters EF; ERS Rehabilitation and Chronic Care, and Physiotherapists Scientific Groups; American Association of Cardiovascular and Pulmonary Rehabilitation; ATS Pulmonary Rehabilitation Assembly and the ERS COPD Audit team. Differences in content and organisational aspects of pulmonary rehabilitation programmes. Eur Respir J. 2014 May;43(5):1326-37. doi: 10.1183/09031936.00145613. Epub 2013 Dec 12. PMID 24337043
- [Background] Casaburi R, Patessio A, Ioli F, Zanaboni S, Donner CF, Wasserman K. Reductions in exercise lactic acidosis and ventilation as a result of exercise training in patients with obstructive lung disease. Am Rev Respir Dis. 1991 Jan;143(1):9-18. doi: 10.1164/ajrccm/143.1.9. PMID 1986689
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Vogiatzis I, Nanas S, Roussos C. Interval training as an alternative modality to continuous exercise in patients with COPD. Eur Respir J. 2002 Jul;20(1):12-9. doi: 10.1183/09031936.02.01152001. PMID 12166558
- [Background] Beauchamp MK, Nonoyama M, Goldstein RS, Hill K, Dolmage TE, Mathur S, Brooks D. Interval versus continuous training in individuals with chronic obstructive pulmonary disease--a systematic review. Thorax. 2010 Feb;65(2):157-64. doi: 10.1136/thx.2009.123000. Epub 2009 Dec 8. PMID 19996334
- [Background] Morris NR, Walsh J, Adams L, Alision J. Exercise training in COPD: What is it about intensity? Respirology. 2016 Oct;21(7):1185-92. doi: 10.1111/resp.12864. PMID 27623321
- [Background] Zoladz JA, Korzeniewski B. Physiological background of the change point in VO2 and the slow component of oxygen uptake kinetics. J Physiol Pharmacol. 2001 Jun;52(2):167-84. PMID 11453098
- [Background] Vogiatzis I, Simoes DC, Stratakos G, Kourepini E, Terzis G, Manta P, Athanasopoulos D, Roussos C, Wagner PD, Zakynthinos S. Effect of pulmonary rehabilitation on muscle remodelling in cachectic patients with COPD. Eur Respir J. 2010 Aug;36(2):301-10. doi: 10.1183/09031936.00112909. Epub 2010 Jan 28. PMID 20110400
- [Background] Hodson M, Sherrington R. Treating patients with chronic obstructive pulmonary disease. Nurs Stand. 2014 Nov 4;29(9):50-8. doi: 10.7748/ns.29.9.50.e9061. PMID 25351094
- [Background] Revill SM, Morgan MD, Singh SJ, Williams J, Hardman AE. The endurance shuttle walk: a new field test for the assessment of endurance capacity in chronic obstructive pulmonary disease. Thorax. 1999 Mar;54(3):213-22. doi: 10.1136/thx.54.3.213. PMID 10325896
- [Background] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Background] Eaton T, Young P, Nicol K, Kolbe J. The endurance shuttle walking test: a responsive measure in pulmonary rehabilitation for COPD patients. Chron Respir Dis. 2006;3(1):3-9. doi: 10.1191/1479972306cd077oa. PMID 16509172
- [Background] Hill K, Dolmage TE, Woon L, Coutts D, Goldstein R, Brooks D. A simple method to derive speed for the endurance shuttle walk test. Respir Med. 2012 Dec;106(12):1665-70. doi: 10.1016/j.rmed.2012.08.011. Epub 2012 Sep 8. PMID 22967491
- [Background] Pepin V, Brodeur J, Lacasse Y, Milot J, Leblanc P, Whittom F, Maltais F. Six-minute walking versus shuttle walking: responsiveness to bronchodilation in chronic obstructive pulmonary disease. Thorax. 2007 Apr;62(4):291-8. doi: 10.1136/thx.2006.065540. Epub 2006 Nov 10. PMID 17099077
- [Background] Borel B, Pepin V, Mahler DA, Nadreau E, Maltais F. Prospective validation of the endurance shuttle walking test in the context of bronchodilation in COPD. Eur Respir J. 2014 Nov;44(5):1166-76. doi: 10.1183/09031936.00024314. Epub 2014 Sep 3. PMID 25186261
- [Background] Demeyer H, Louvaris Z, Frei A, Rabinovich RA, de Jong C, Gimeno-Santos E, Loeckx M, Buttery SC, Rubio N, Van der Molen T, Hopkinson NS, Vogiatzis I, Puhan MA, Garcia-Aymerich J, Polkey MI, Troosters T; Mr Papp PROactive study group and the PROactive consortium. Physical activity is increased by a 12-week semiautomated telecoaching programme in patients with COPD: a multicentre randomised controlled trial. Thorax. 2017 May;72(5):415-423. doi: 10.1136/thoraxjnl-2016-209026. Epub 2017 Jan 30. PMID 28137918